CLINICAL TRIAL: NCT00914173
Title: A Single-blind Randomized Clinical Trial to Assess the Efficacy of the Medasense's Non-Invasive Pain Monitor in Estimating the Pain Level Comparing to the Pain Stimuli and the Reported Pain Level on Healthy Subjects.
Brief Title: Pain Monitoring Using Plurality of Non-invasive Physiological Measurement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medasense Biometrics Ltd (Other)
Responsible Party: Elon Eisenberg, MD, Rambam medical Center -The Pain palliation unit
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: Medasense001
Record Dates: First submitted 2009-06-03; First posted 2009-06-04 (Estimated); Last update posted 2010-01-28 (Estimated); Status verified 2010-01

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pain/No Pain Stimuli (Experimental): One Arm is used in this trial. The comparator is within the arm. The different types of stimuli levels and types are compared.
  Interventions: Device: Scanlaf Circulator and water bath; Device: Medoc TSA 2000

INTERVENTIONS:
Device: Scanlaf Circulator and water bath — Cold Pressor Test
  Other Names: Open Cold Water Bath
Device: Medoc TSA 2000 — Thermal stimuli pain
  Other Names: Medoc Advanced Medical Systems TSA-II System

SUMMARY:
The clinical trial is intended to implement, validate performances and evaluate efficacy of the pain monitoring device for automated assessment of patient's pain level. The efficacy of the pain monitor will be tested by comparing its results to the patient pain reports towards a given pain stimuli.

DETAILED DESCRIPTION:
Pain is an unpleasant sensation, ranging from slight discomfort to intense suffering. However, since a great extent of pain is a subjective phenomenon, it has frequently defied objective, quantitative measurement. Traditionally, physicians have had to assess a patient's pain by relying on the patient's own description. Self-description is not only subjective by definition; it is often inaccurate, in part because it is difficult for subjects to precisely articulate their pain while in the midst of a pain experience. Moreover, the report might be impossible when the subject cannot communicate

Presently, in order to quantify pain, the care provider asks the patient to rate his/her pain intensity using one-dimensional scale usually scored from 0 to 10. This scale is known as Numeric Pain Scale. This and other measures are used by the care providers to estimate the correct treatment dose and or to track a treatment progress. Due to its impact on care provider decision to prescribe painkiller mediation, some patients also intentionally misrepresent the existence or extent of their pain. Yet, without any reliable basis for denying such prescriptions, physicians generally must assume that the claims are truthful, even when they may suspect a lack of sincerity. Otherwise, the care provider may be accused of inhumane treatment. Conversely, other patients may underreport their pain, again for a variety of reasons.

The presented clinical trial is intended to implement, validate performances and evaluate efficacy of the pain monitoring device for automated assessment of patient's pain level. During the trial, up to 100 healthy young adults will be voluntarily inflicted by pain stimuli. The pain stimuli will be thermal heat pain stimulus and cold water pain stimulus applied with different intensities. Plurality of Non-Invasive Physiological Measurements will be recorded from volunteers and their Numeric Pain Scale reports will be monitored before, during and after the pain induction. Additional information such as age, gender, ethnicity, etc. will be collected as well. The collected database will be used to implement the algorithm that applies modern signal processing and machine learning methods in order to differentiate between different pain levels. The algorithm will be later integrated into pain monitoring device. The efficacy of the algorithm of the pain monitor will be tested by comparing its results to the patient pain reports towards a given pain stimuli.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participant that response to pain stimuli
* Blood Pressure < (90,140), Heart Rate < 100pps
* Patient informed consent must be obtained

Exclusion Criteria:

* Not responding to pain stimuli (Hypoalgesia)
* Over responding to pain stimuli (Hyperalgesia)
* Classifying non pain stimuli as painful event (Allodynia)
* Medication/drugs were taken in the last week
* Usage of chronic medication in the last 3 months (not including contraceptive pills)
* Alcohol usage during the last 48 hours
* Caffeine in the last 3 hours
* Pregnant women
* Inability to comply with the study protocol.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Comparison between the pain monitoring device results and the subjective pain report measured by the numeric pain scale to a given pain stimulus (heat and cold) | one year

SECONDARY OUTCOMES:
Collect database to implement the algorithm for the pain monitor to differ between different pain levels. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Elon Eisenberg, Prof., Principal Investigator — Pain Relief Unit, Rambam Health Care Campus
Locations (1):
- Pain Relief Unit,Rambam Medical Center, Haifa, Israel